CLINICAL TRIAL: NCT06688188
Title: 68Ga-JH12 PET/CT: Dosimetry and Biodistribution Study in Patients With Various Cancers
Brief Title: 68Ga-JH12 PET/CT: Dosimetry and Biodistribution Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-JH12
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dynamic PET scans (Experimental): PET imaging will begin at 3 minutes, 15 minutes, 30min minutes, 60 minutes and 150 minutes after injection.
  Interventions: Drug: 68Ga-JH12

INTERVENTIONS:
Drug: 68Ga-JH12 — The dose will be 148-222 MBq given intravenously.

SUMMARY:
68Ga-JH12 is a novel radiotracer targeting C-X-C motif chemokine receptor 4 (CXCR4). In this study, we observed the safety, biodistribution, and radiation dosimetry of 68Ga-JH12 in patients with different types of cancer.

DETAILED DESCRIPTION:
C-X-C motif chemokine receptor 4 (CXCR4) is highly expressed in patients affected with malignant tumors and ex-vivo analyses provided evidence that the expression level on the tumor cell surface is tightly linked to the proliferation index. In recent years, the diagnostic PET agent 68Ga-Pentixafor targeting this chemokine receptor has been extensively validated in haematological malignancies and solid tumors. 68Ga-JH12, a novel radiopharmaceutical targeting CXCR4, demostrated high stability in vitro and in vivo, and can accumulate specifically in tumors with high binding affinity, safety, and selectivity in preclinical studies. In this study, the safety, biodistribution, and radiation dosimetry of 68Ga-JH12 in patients with Various Cancers were observed to evaluate the dosimetric characteristics of 68Ga-JH12.

ELIGIBILITY:
Inclusion Criteria:

* Various solid tumors with available histopathological findings
* Signed informed consent

Exclusion Criteria:

* pregnant or lactational women
* who suffered from severe hepatic and renal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | up to 1 week
  Hematologic status, liver function, renal function and General vital signs were recorded before and 1 week after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Dosimetry of normal organs and tumors | From right after tracer injection to 150 minutes at post-injection
  The semiquantitative dosimetry will be performed based on PET/CT acquisitions after the first administration of 68Ga-JH12. The dose delivered to normal organs and tumors will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China